CLINICAL TRIAL: NCT04881591
Title: Improving Adherence and Safety of Orthopedic Treatment of Idiopathic Scoliosis in Adolescents Using Information and Communication Technologies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ScoliosisAPP
Record Dates: First submitted 2021-04-07; First posted 2021-05-11 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence; Brace
Keywords: ICT; Treatment Adherence; Treatment efficacy; Treatment safety
MeSH Terms: conditions — Scoliosis; Treatment Adherence and Compliance | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: One condition
Masking Description: Patients will be informed of the condition they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APP+Usual Treatment (Experimental): Participants at this condition will receive the usual medical treatment for their scoliosis but also they will be monitored daily using the Scoliosis Pain Monitor APP. Alarms will be generated in the face of certain preestablished undesired events. Physicians will be asked to call patients and change/stop treatment if an alarm is received.
  Interventions: Device: Treatment as usual + APP

INTERVENTIONS:
Device: Treatment as usual + APP — Participants at this condition will receive the usual medical treatment for their scoliosis but also they will be monitored daily using the Scoliosis Pain Monitor APP. Alarms will be generated in the face of certain preestablished undesired events. Physicians will be asked to call patients and change/stop treatment if an alarm is received.

SUMMARY:
The present project aims to test the feasibility of a new management mechanism for inter-visit monitoring of adolescent patients with idiopathic scoliosis that improves the quality and safety of current orthopedic treatments using information and communication technologies (ICT).

DETAILED DESCRIPTION:
Idiopathic scoliosis is defined as a spinal deformity affecting the anteroposterior plane and exceeding 10 degrees of angulation. The label idiopathic arises from ruling out other causes, such as tumors, trauma or infections, that may explain the deformity. This pathology affects approximately 2% of the population, being up to 5 times more frequent in girls than in boys and age playing a fundamental role in the progression and worsening of the problem.

In most cases, scoliosis appears during adolescence (up to 89% of cases according to studies), being very rare up to 3 years of age (between 1% and 5% of detected cases) and slightly more frequent in the infantile stage (7 to 10.5% of scoliosis cases). Scoliosis often does not cause pain or other complications associated with the deformity. However, as the curvature deformity increases (especially after 25 degrees), complications become more pronounced and treatment becomes necessary. For example, in the case of curvatures between 30 and 40 degrees and curves between 20 and 29 degrees that have progressed rapidly in the last year (more than 5 degrees), bracing has become the indicated treatment, while more invasive intervention (surgery) will be necessary in more severe cases.

The prevalence of cases requiring treatment (by bracing or, in the worst case, surgery) is estimated to be between 0.2 and 0.3% of the population under 18 years of age. However, although in many cases scoliosis is not associated with medical complications, it has been shown that, even in people with less severe curvature, this deformity is associated with psychological complications, such as lower self-esteem, a more depressed mood, high alcohol consumption and even suicidal ideation, which are aggravated during treatment.

Through bracing, applied early on, it is hoped that the proper curvature of the spine will be aided by the guidance imposed by the brace. However, although review studies indicate promising results with this intervention, they also indicate that the use of bracing does not yet possess sufficient scientific evidence. This is mainly due, as indicated by the literature, to the low adherence to bracing in this population, which tends to be exaggerated when evaluated retrospectively. Given that one of the best predictors of the effectiveness of orthopedic treatment of scoliosis is, in fact, time in brace use, greater efforts should be made to improve adherence to treatment in this population. Some authors have proposed that factors such as beliefs about the pathology and treatment (e.g., "I don't care about my back" or "I think people will see the brace under my clothes"), as well as the undesirable effects of brace use (e.g., chafing, discomfort when sleeping, or pain), may be at least partly responsible for this low adherence.

With the aforementioned purpose in mind, we hope that the use of our Pain Monitor App, which has been recently validated in an empirical study, will allow early detection of low adherence to brace use, the appearance of undesirable effects of its use or the persistence of dysfunctional beliefs. All this with the aim of acting quickly to promote their adherence to brace use, make changes to the brace when it causes undesirable effects, or perform psychoeducational interventions when dysfunctional beliefs about scoliosis or treatment persist. As a result of the above, we expect to increase the effectiveness of the intervention (better curvature evolution) and the quality of life and emotional well-being of the patients. Avoiding progression of the curvature is important since surgery is associated with significant post-surgical complications, such as infections and mechanical and neurological problems, with low success rate and frequent need for several surgeries, while untreated scoliosis in the adult is often accompanied by chronic low back pain and significant instability.

ELIGIBILITY:
Inclusion Criteria:

* Adolescente patient (between 10 and 18 years old)
* Wearing a brace for less than 3 months
* The patient has a mobile phone with Android or iOS operating systems
* The patients has the physical ability to use the application
* The patient does not present psychological and or cognitive alterations/ problems with language that make their participation difficult
* The patient (or the legal tutor) voluntarily wants to participate and sings the informed consent

Exclusion Criteria:

* The patient does not have an own mobile phone or has a mobile phone with uncompatible characteristics
* Cognitive alterations, lenguage problems to understand the use of the app and to respond its questions
* The patient presents a severe mental health issues or substance abuse.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
App' usability will be assessed by the SUS | During the app use (one week after app first use)
  The System Usability Scale will be administered to assess the perception that a tool is simple to use and useful. It is composed by 10 items which are responded according to a 5-point Likert scale (1 = "completely disagree" to 5 ="completely agree"). Half of the items are recorded so that higher scores in the scale represent higher usability. Total scores are converted into percentages from 0% to 100%.
App' usability will be assessed by the SUS | Immediately after the app use (3 months after app first use)
  The System Usability Scale will be administered to assess the perception that a tool is simple to use and useful. It is composed by 10 items which are responded according to a 5-point Likert scale (1 = "completely disagree" to 5 ="completely agree"). Half of the items are recorded so that higher scores in the scale represent higer usability. Total scores are converted into percentages from 0% to 100%.
App' acceptability will be assessed by the SUS | During the app use (one week after app first use)
  The System Usability Scale will be administered to assess the perception that a tool is simple to use and useful. It is composed by 10 items which are responded according to a 5-point Likert scale (1 = "completely disagree" to 5 ="completely agree"). Half of the items are recorded so that higher scores in the scale represent higer usability. Total scores are converted into percentages from 0% to 100%.
App' acceptability will be assessed by the SUS | Immediately after the app use (3 months after app first use)
  The System Usability Scale will be administered to assess the perception that a tool is simple to use and useful. It is composed by 10 items which are responded according to a 5-point Likert scale (1 = "completely disagree" to 5 ="completely agree"). Half of the items are recorded so that higher scores in the scale represent higer usability. Total scores are converted into percentages from 0% to 100%.
Feasibility of the study will be assessed by a calculation of responses completed | Immediately after the app use (3 months after app first use)
  Percentage of completed assessments in the app compared to the number of planned evaluations will be calculated

SECONDARY OUTCOMES:
Stress | Twice: at baseline (beggining of the study, before the brace use) and at end of the study (3 months after app first use)
  It will be measured with the Sobberheim Stress Questionnaire (BSSQ brace). It contains 8 items responded based on a 4-points Likert scale (0= "most stress" to 3 = "least stress"). Total scores range from 0 to 24, higher total scores indicating lower stress.
Patients' Quality of life | Twice: at baseline (beggining of the study, before the brace use) and at end of the study (3 months after app first use)
  It will be measured with the Italian Spine Youth Quality Of Life (ISYQOL). It is composed by 20 items responded by a 3-points Likert scale (0= "never"; 1 = "sometimes"; 2= "often").Total scores are converted into percentages from 0% to 100%, higher percentages indicating greater quality of life.
Perceived health status | Twice: at baseline (beggining of the study, before the brace use) and at end of the study (3 months after app first use)
  It will be measured with the Scoliosis Research Society -22 (SRS-22). It is composed by 22 items, response rate range from 1= "Severe" to 5= "None". Total score range from 22 to 110, higher scores indicating greater perceived health status.
Anxiety and depressive symptoms | Twice: at baseline (beggining of the study, before the brace use) and at end of the study (3 months after app first use)
  It will be measured with the Hospital Anxiety and Depression Scale (HADS). It consists of 14 items. Each item is rated according to a 4-point Likert scale from 0= "as much as I always do" to 3 = "not at all". Total scores range between 0 and 21, higher scores represent higher anxiety and depressive symptoms.
Mood | Daily up to 3 months
  Questions adapted and validated from the Profile of Mood States and Short Form 12
Brace adherence | Daily up to 3 months
  Adherence will be calculated by dividing the number of hours of use reported and the prescription filled
Treatment safety: Brace-related side effects | Daily up to 3 months
  An ad hoc question will be created including the most frequent side effects according to the literature and to professionals clinical expertise

CONTACTS AND LOCATIONS:
Overall Officials: Azucena García-Palacios, PhD, Study Chair — Universitat Jaume I; Judith Sánchez-Raya, PhD, Study Chair — Hospitla Universitario Vall d'Hebron; Amanda Díaz-García, PhD, Study Chair — Universidad de Zaragoza; Diana Castilla, PhD, Study Chair — University of Valencia; Verónica Martínez-Borba, MsC, Study Chair — Universitat Jaume I
Locations (1):
- Vall d'Hebron Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Only Dra. Sánchez-Raya will be able to access to individual participant data.

REFERENCES:
- [Background] Aebi M. The adult scoliosis. Eur Spine J. 2005 Dec;14(10):925-48. doi: 10.1007/s00586-005-1053-9. Epub 2005 Nov 18. PMID 16328223
- [Background] Charosky S, Guigui P, Blamoutier A, Roussouly P, Chopin D; Study Group on Scoliosis. Complications and risk factors of primary adult scoliosis surgery: a multicenter study of 306 patients. Spine (Phila Pa 1976). 2012 Apr 15;37(8):693-700. doi: 10.1097/BRS.0b013e31822ff5c1. PMID 22504517
- [Background] D'Astous JL, Sanders JO. Casting and traction treatment methods for scoliosis. Orthop Clin North Am. 2007 Oct;38(4):477-84, v. doi: 10.1016/j.ocl.2007.03.006. PMID 17945127
- [Background] Dunn J, Henrikson NB, Morrison CC, Blasi PR, Nguyen M, Lin JS. Screening for Adolescent Idiopathic Scoliosis: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Jan 9;319(2):173-187. doi: 10.1001/jama.2017.11669. PMID 29318283
- [Background] Fong DY, Lee CF, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Luk KD. A meta-analysis of the clinical effectiveness of school scoliosis screening. Spine (Phila Pa 1976). 2010 May 1;35(10):1061-71. doi: 10.1097/BRS.0b013e3181bcc835. PMID 20393399
- [Background] Janicki JA, Alman B. Scoliosis: Review of diagnosis and treatment. Paediatr Child Health. 2007 Nov;12(9):771-6. doi: 10.1093/pch/12.9.771. PMID 19030463
- [Background] Lenssinck ML, Frijlink AC, Berger MY, Bierman-Zeinstra SM, Verkerk K, Verhagen AP. Effect of bracing and other conservative interventions in the treatment of idiopathic scoliosis in adolescents: a systematic review of clinical trials. Phys Ther. 2005 Dec;85(12):1329-39. PMID 16305271
- [Background] Morton A, Riddle R, Buchanan R, Katz D, Birch J. Accuracy in the prediction and estimation of adherence to bracewear before and during treatment of adolescent idiopathic scoliosis. J Pediatr Orthop. 2008 Apr-May;28(3):336-41. doi: 10.1097/BPO.0b013e318168d154. PMID 18362800
- [Background] Negrini S, Atanasio S, Zaina F, Romano M. Rehabilitation of adolescent idiopathic scoliosis: results of exercises and bracing from a series of clinical studies. Europa Medicophysica-SIMFER 2007 Award Winner. Eur J Phys Rehabil Med. 2008 Jun;44(2):169-76. PMID 18418337
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Reichel D, Schanz J. Developmental psychological aspects of scoliosis treatment. Pediatr Rehabil. 2003 Jul-Dec;6(3-4):221-5. doi: 10.1080/13638490310001644593. PMID 14713589
- [Background] Suso-Ribera C, Castilla D, Zaragoza I, Ribera-Canudas MV, Botella C, Garcia-Palacios A. Validity, Reliability, Feasibility, and Usefulness of Pain Monitor: A Multidimensional Smartphone App for Daily Monitoring of Adults With Heterogenous Chronic Pain. Clin J Pain. 2018 Oct;34(10):900-908. doi: 10.1097/AJP.0000000000000618. PMID 29659375
- [Background] Tones M, Moss N, Polly DW Jr. A review of quality of life and psychosocial issues in scoliosis. Spine (Phila Pa 1976). 2006 Dec 15;31(26):3027-38. doi: 10.1097/01.brs.0000249555.87601.fc. PMID 17173000
- [Background] Weinstein SL, Dolan LA, Cheng JC, Danielsson A, Morcuende JA. Adolescent idiopathic scoliosis. Lancet. 2008 May 3;371(9623):1527-37. doi: 10.1016/S0140-6736(08)60658-3. PMID 18456103
- [Background] Yaman O, Dalbayrak S. Idiopathic scoliosis. Turk Neurosurg. 2014;24(5):646-57. doi: 10.5137/1019-5149.JTN.8838-13.0. PMID 25269032
- [Background] Yang S, Andras LM, Redding GJ, Skaggs DL. Early-Onset Scoliosis: A Review of History, Current Treatment, and Future Directions. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-0709. Epub 2015 Dec 7. PMID 26644484